CLINICAL TRIAL: NCT01556204
Title: Laparoscopy vs. Robotic Surgery for Endometriosis (LAROSE): a Prospective Randomized Controlled Trial
Acronym: LAROSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12-173
Record Dates: First submitted 2012-03-13; First posted 2012-03-16 (Estimated); Results first posted 2016-08-04 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2016-12

CONDITIONS: Endometriosis
Keywords: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Robotic Surgical Procedures; Laparoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Robotic Surgery (Experimental): Robotic surgery using the da Vinci Surgical System
  Interventions: Procedure: Robotic surgery
- Laparoscopy (Active Comparator): Laparoscopic assisted resection of endometriosis will be performed using up to five 5mm ports.
  Interventions: Procedure: Laparoscopic Surgery

INTERVENTIONS:
Procedure: Robotic surgery — The technique for resection of superficial and deep endometriosis will be performed in a standard fashion. All superficial lesions suspicious for endometriosis (pigmented and non-pigmented) will be completely resected until non-diseased peritoneal margins are visualized around the defect or will be fulgurized using bipolar energy; all deep lesions suspicious for endometriosis will be completely resected until non-diseased margins are visualized in the tissue surrounding the defect. Cystectomy(ies) will be performed for endometrioma(s). The fascia of any port greater or equal to 10mm will be reapproximated. Cystoscopy would only be performed when deemed appropriate by the surgeon (e.g., to assess for lower urinary tract injury in cases that require extensive ureterolysis).
  Arms: Robotic Surgery
Procedure: Laparoscopic Surgery — The technique for resection of superficial and deep endometriosis will be performed in a standard fashion. All superficial lesions suspicious for endometriosis (pigmented and non-pigmented) will be completely resected until non-diseased peritoneal margins are visualized around the defect or will be fulgurized using bipolar energy; all deep lesions suspicious for endometriosis will be completely resected until non-diseased margins are visualized in the tissue surrounding the defect. Cystectomy(ies) will be performed for endometrioma(s). The fascia of any port greater or equal to 10mm will be reapproximated. Cystoscopy would only be performed when deemed appropriate by the surgeon (e.g., to assess for lower urinary tract injury in cases that require extensive ureterolysis).
  Other Names: Laparoscopy
  Arms: Laparoscopy

SUMMARY:
The objective of this study is to conduct a prospective randomized controlled trial of robotic-assisted versus conventional laparoscopy for the treatment of endometriosis.

DETAILED DESCRIPTION:
This is a prospective randomized control trial. Study subjects will be recruited from patients that present to the Department of Gynecology who are to have surgery for endometriosis at the Cleveland Clinic.

Patient that require bowel resection and/or ureteral reanastomosis are not included due to the fact that these events impact operating time significantly and are not commonly performed as part of endometriosis surgery (subjects may not be equally distributed among both arms).

Eligible patients that agree to participate will be provided written informed consent administered by the collaborators listed on this Institutional Review Board (IRB) at the above clinic locations. In addition to a standardized evaluation including the history and physical examination, the patients will complete the validated health-related quality of life questionnaires SF-12 and Endometriosis Health Profile-30 (EHP-30) with additional questions to determine baseline pain and activity scales as well as daily pain medication use.

Surgeries will be performed by two board certified gynecologic surgeons (TF and JG). JG will participate in the laparoscopic arm of the study (Beachwood Family Health and Surgery Center) while TF will participate in both arms (Cleveland Clinic main campus). The patients of JG randomized to robotic surgery will be performed by TF at Cleveland Clinic main campus.

Additionally, after the surgery, the patients will complete the above questionnaires as well as diaries addressing narcotic use and quality of life at 6 weeks and 6 months. Completion of questionnaires and diaries is the only additional assessment that is specific to participation in this study that is not usually included as part of the standard care for the treatment of endometriosis. It should take no more than 10 minutes to complete the questionnaires and less than 5 minutes each day to complete the diaries. The study subjects will not be exposed to any additional risk by participating in this study except for the inconvenience of completing the questionnaires and daily diaries.

The participants will be randomized preoperatively (at the time of surgery scheduling) according to a computer-generated randomization schedule with random block sizes with the use of the SAS statistical software package (SAS Institute, Cary, NC). All patients will be blinded to their assignment. Intraoperative randomization of the patients is not feasible due to the fact that the operating room staff and operating room assigned for a given case is different for robotic and traditional laparoscopic cases.

Patients who do not choose to participate in this study will still be offered the standard evaluation and management including laparoscopic treatment of endometriosis as deemed appropriate by the primary surgeon. Robotic-assisted laparoscopic treatment of endometriosis is not routinely performed in this institution however, and thus is not considered part of the standard of care.

Laparoscopic assisted resection of endometriosis will be performed using up to five 5mm. ports. An umbilical port will be placed for the laparoscope and additional ports as dictated by each individual surgery. The robotic-assisted resection of endometriosis will be performed using the da Vinci Surgical System (Intuitive Surgical Inc., Sunnyvale, CA, USA) using up to five ports as needed. An umbilical port will be placed for the laparoscope (10/12mm), a 5mm assistant port will be placed in the right lower quadrant and two or three 8 mm robotic ports will be placed in the lower quadrants bilaterally.

The technique for resection of superficial and deep endometriosis will be performed in a standard fashion. All superficial lesions suspicious for endometriosis (pigmented and non-pigmented) will be completely resected until non-diseased peritoneal margins are visualized around the defect or will be fulgurized using bipolar energy; all deep lesions suspicious for endometriosis will be completely resected until non-diseased margins are visualized in the tissue surrounding the defect. Cystectomy(ies) will be performed for endometrioma(s). The fascia of any port greater or equal to 10mm will be reapproximated. Cystoscopy would only be performed when deemed appropriate by the surgeon (e.g., to assess for lower urinary tract injury in cases that require extensive ureterolysis).

Patients that are found not to have endometriosis at the time of surgery will be excluded from the study. The robot will be docked for all cases assigned for this arm irrespective of the amount of disease encountered (including mild endometriosis).

Data points recorded during the procedure will include: operating room time of entry and exit and time from incision to closure. From this information, the operating room costs and anesthesia costs, i.e., the amount that a provider must pay for goods or services, will be calculated. Estimated blood loss, perioperative and post-operative complications, and number of days in the hospital (in cases that warrant admission) will be calculated. The standard American Society of Reproductive Medicine (ASRM) intraoperative endometriosis scoring system will be documented at the end of each surgery. Procedure and inpatient hospital costs (if applicable) will also be determined. All the operating room data (including the primary outcome) will be collected by a research nurse or coordinator that will be assigned for this task (to optimize reliability of these measurements).

Patients will complete their daily narcotic use, which will include oral as well as patient-controlled analgesia IV narcotic use in the hospital when applicable as well as quality of life diaries. Patients will return to clinic for a two week post-operative visit.

Prior to surgery, the patients will undergo a physical examination by a physician who is blinded to the patient's surgical group assignments. Additionally, patients will fill out the SF-12 health survey, EHP-30 and activity assessment questionnaires, pain scale and daily pain medication / narcotic use at baseline.

At the 2 week postoperative visit, a routine physical exam will be performed, the daily pain medication diary will be retrieved and the questionnaires for surgical pain and activity assessment will be applied.

At 6 weeks and 6 months, the nurse or physician will repeat the questionnaires by email (using Redcap), mailed questionnaires or over the telephone (SF-12, EHP-30, pain scales, daily pain medication / narcotic use and activity assessment questionnaires). The physician or nurse will also collect all the intraoperative and inpatient data for this project as well as review the medical record for possible admissions and postoperative complications.

All data points and demographic information will be recorded in a secured, password protected database on the Gynresearch drive that will only be assessed by the collaborators on this IRB. Subjects will only be identified by their Cleveland Clinic medical record number. It is necessary to identify patients in this manner so that their clinical progress (e.g. postoperative complications, emergency room visits) can be located and recorded on the database.

ELIGIBILITY:
Inclusion Criteria:

* women 18 years of age or greater who are to undergo laparoscopic treatment of presumed endometriosis, as determined clinically by the operating surgeon.

Exclusion Criteria:

* suspected malignancy,
* medical illness precluding laparoscopy,
* inability to give informed consent,
* morbid obesity (BMI > 44), or
* need for concomitant bowel resection and/or ureteral reanastomosis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2012-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tommaso Falcone, MD, Principal Investigator — The Cleveland Clinic
Locations (3):
- United States (3):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Soto E, Luu TH, Liu X, Magrina JF, Wasson MN, Einarsson JI, Cohen SL, Falcone T. Laparoscopy vs. Robotic Surgery for Endometriosis (LAROSE): a multicenter, randomized, controlled trial. Fertil Steril. 2017 Apr;107(4):996-1002.e3. doi: 10.1016/j.fertnstert.2016.12.033. Epub 2017 Feb 24. PMID 28238489

RESULTS

PARTICIPANT FLOW:
Groups:
- Robotic Surgery: da Vinci Surgical System
  Surgery for endometriosis: The technique for resection of superficial and deep endometriosis will be performed in a standard fashion. All superficial lesions suspicious for endometriosis (pigmented and non-pigmented) will be completely resected until non-diseased peritoneal margins are visualized around the defect; all deep lesions suspicious for endometriosis will be completely resected until non-diseased margins are visualized in the tissue surrounding the defect. Cystectomy(ies) will be performed for endometrioma(s). The fascia of any port greater or equal to 10mm will be reapproximated. Cystoscopy would only be performed when deemed appropriate by the surgeon (e.g., to assess for lower urinary tract injury in cases that require extensive ureterolysis).
- Laparoscopy: Laparoscopic assisted resection of endometriosis will be performed using up to five 5mm ports.
  Surgery for endometriosis: The technique for resection of superficial and deep endometriosis will be performed in a standard fashion. All superficial lesions suspicious for endometriosis (pigmented and non-pigmented) will be completely resected until non-diseased peritoneal margins are visualized around the defect; all deep lesions suspicious for endometriosis will be completely resected until non-diseased margins are visualized in the tissue surrounding the defect. Cystectomy(ies) will be performed for endometrioma(s). The fascia of any port greater or equal to 10mm will be reapproximated. Cystoscopy would only be performed when deemed appropriate by the surgeon (e.g., to assess for lower urinary tract injury in cases that require extensive ureterolysis).
Period: Overall Study
Arm/Group | Robotic Surgery | Laparoscopy
Started | 35 | 38
Completed | 35 | 38
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Robotic: Robotic surgery
- Laparoscopic: Laparoscopic surgery
- Total: Total of all reporting groups
Arm/Group | Robotic | Laparoscopic | Total
Number analyzed (Participants) | 35 | 38 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.3 (7.2) | 34.5 (8.5) | 34.5 (8.5)
Gender [Count of Participants; unit: Participants]
  Female | 35 | 38 | 73
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 35 | 38 | 73

OUTCOME MEASURES:

1. Primary Outcome: Operative Time
Description: Operative time is defined as skin incision to skin closure.
Time Frame: 1st 24 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Robotic Surgery | Laparoscopy
Number analyzed (Participants) | 35 | 38
minutes | 106.6 (48.8) | 101.6 (63.2)
Statistical Analysis 1: Comparison: Robotic Surgery vs Laparoscopy; Variance estimates for this power analysis were taken from Nezhat C, et al, 2010. We determined that 37 subjects in each arm were needed to detect a difference of ≥ 32 minutes in operating time between conventional and robotic surgery for endometriosis with 80% power and a significance level of 0.05; Test type: Superiority or Other; p = 0.71, t-test, 2 sided — This p-value is from a single comparison between two arms for operative time

2. Secondary Outcome: Pain
Description: Pain as estimated by endometriosis, Endometriosis Health Profile-30 (EHP-30). Score ranges from 0-100. Lower score denotes improvement. Pain: As score decreases, pain decreases. No subscales.
Time Frame: Baseline, 6-weeks, 6-months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Robotic Surgery | Laparoscopy
Number analyzed (Participants) | 35 | 38
units on a scale
  Baseline | 51.2 (18.1) | 54.2 (16)
  6-weeks | 28.6 (23.7) | 25.3 (21.6)
  6-months | 24.8 (26.5) | 21.5 (23.9)
Statistical Analysis 1: Comparison: Robotic Surgery vs Laparoscopy; Secondary analysis for pain at baseline for robotic vs conventional laparoscopy for endometriosis; Test type: Superiority or Other; p = 0.53, Mixed Models Analysis — This applies to Row title: Baseline
Statistical Analysis 2: Comparison: Robotic Surgery vs Laparoscopy; Pain scores at 6 weeks comparison between robotic and laparoscopy; Test type: Superiority or Other; p = 0.53, Mixed Models Analysis — This applies to Row title: 6-weeks
Statistical Analysis 3: Comparison: Robotic Surgery vs Laparoscopy; Pain scores at 6 months for robotic vs laparoscopy; Test type: Superiority or Other; p = 0.48, Mixed Models Analysis — This applies to Row title: 6-months

ADVERSE EVENTS:
Groups:
- Robotic Surgery: da Vinci Surgical System
  Surgery for endometriosis: The technique for resection of superficial and deep endometriosis will be performed in a standard fashion. All superficial lesions suspicious for endometriosis (pigmented and non-pigmented) will be completely resected until non-diseased peritoneal margins are visualized around the defect or will be fulgurized using bipolar energy; all deep lesions suspicious for endometriosis will be completely resected until non-diseased margins are visualized in the tissue surrounding the defect. Cystectomy(ies) will be performed for endometrioma(s). The fascia of any port greater or equal to 10mm will be reapproximated. Cystoscopy would only be performed when deemed appropriate by the surgeon (e.g., to assess for lower urinary tract injury in cases that require extensive ureterolysis).
- Laparoscopy: Laparoscopic assisted resection of endometriosis will be performed using up to five 5mm ports.
  Surgery for endometriosis: The technique for resection of superficial and deep endometriosis will be performed in a standard fashion. All superficial lesions suspicious for endometriosis (pigmented and non-pigmented) will be completely resected until non-diseased peritoneal margins are visualized around the defect or will be fulgurized using bipolar energy; all deep lesions suspicious for endometriosis will be completely resected until non-diseased margins are visualized in the tissue surrounding the defect. Cystectomy(ies) will be performed for endometrioma(s). The fascia of any port greater or equal to 10mm will be reapproximated. Cystoscopy would only be performed when deemed appropriate by the surgeon (e.g., to assess for lower urinary tract injury in cases that require extensive ureterolysis).
Arm/Group | Robotic Surgery | Laparoscopy
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/38
Other Adverse Events (participants affected / at risk) | 0/35 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes